CLINICAL TRIAL: NCT04167566
Title: Exploring the Impact of Scaling up Mass Testing, Treatment and Tracking on Malaria Prevalence Among Children in the Pakro Sub District of Ghana
Brief Title: Impact of Scaling up Mass Testing, Treatment and Tracking on Malaria Prevalence Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NoguchiMIMR
Record Dates: First submitted 2019-11-05; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Malaria; Malaria, Asymptomatic Parasitaemia
Keywords: Impact; mass testing; treatment; tracking; Malaria prevalence; Children; Pakro Ghana
MeSH Terms: conditions — Malaria; Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: The interventions are designed to compare the baseline to evaluation findings. There are two components to this implementation study a) The longitudinal (cohort) study: This is basically the prevalence surveys to be conducted with the selected cohort of children 6 months to 15 years - at baseline and before each of the subsequent MTTT rounds. b) The Survey involves using structured questionnaire to interview caretakers of children under five to solicit their views on the implementation process perceived benefits and challenges etc. Though the target group is children from 6 months to 15 years of age, all parasitised adults will be cleared of the parasite during the interventions as well to reduce the parasite reservoirs. Prevalence of malaria trends in cohort group over the study period will reveal the effect of MTTT scale-up on the children 6 month to 15 years. Between interventions, the teams will conduct homes-based management of malaria for confirmed febrile cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Communities (Other): All participants confirmed using rapid diagnostic test (RDTs) to be carrying the malaria parasite will be treated using artemisinin combination therapy (ACT) following the Ghana National Malaria Treatment Guidelines and followed up on days 1, 2, 3 during treatment as DOTs (Directly observed therapy) and on day 7 post treatment. The research team together with Community volunteers will be provided the treatment guidelines which specify the dosage for each treatment regimen. Participants who receive the treatment will be observed for five minutes to ensure that they retain the drug. Those who vomit within this period will have the treatment repeated.
  Interventions: Combination Product: Artemisinin Combination Therapy ACTs

INTERVENTIONS:
Combination Product: Artemisinin Combination Therapy ACTs — All participants will be tested using RDTs and all confirmed cases will be treated with ACTs. The ACT regimen use at each time will be the one the National Malaria Control Programme will be using at that particular moment.

SUMMARY:
Malaria poses a serious burden in sub-Sahara Africa. Efforts are ongoing to scale up interventions that work. These include the use of Long Lasting Insecticidal Nets (LLIN), Intermittent Preventive Treatment in children (IPTc), and test, treat and track (TTT). There is the need, however, for mass testing, treatment and tracking (MTTT) of the whole population to reduce the parasite load before implementing the aforementioned interventions. Though, Seasonal Malaria Chemoprophylaxis (SMC) is adopted for selected localities in Ghana, the impact of such interventions could be enhanced, if associated with MTTT in order to reduce the parasite load at baseline. MTTT of children in Ghana has demonstrated a parasite load reduction from 25% to 1%. However, unanswered questions include - could this be scaled up? What proportion of the community could be covered over a given time? What would it take to accomplish large scale MTTT? In designing interventions that aim at reducing the burden of malaria in children under five, for example, MTTT has largely been left out. Adults who are not often targeted by such interventions remain reservoirs that fuel transmission. This study explores the scale-up of interventions that work using existing community volunteer teams to lower cost. These volunteers will play a surveillance role by conducting home-based management of malaria. To avoid challenges posed by stockouts, short message service (SMS) will be used to monitor the level of stocks for malaria medicine and Rapid Diagnostic Tests (RDTs). It is hypothesized that there are more asymptomatic malaria cases (those who carry the parasite but are not ill) than symptomatic cases reported by hospital records in the Pakro sub district and that, carrying out MTTT in combination with home-based management of malaria in specific communities could greatly reduce the burden. Through this study, the bottlenecks that hinder scaling-up of MTTT will be documented in order to facilitate the process.

DETAILED DESCRIPTION:
Introduction/Rationale

The World Health Organization (WHO) in 2010 reported that malaria was endemic in 96 countries reflecting an improvement of the situation of 2005 where it was endemic in 106 countries. Malaria morbidity and mortality remain a serious problem in sub Saharan Africa especially in areas with holo-endemic transmission. Over the last decade, the number of recorded malaria cases has steadily dropped from 247 million cases with 881,000 deaths reported in 2006 to 198 million with 584,000 deaths in 2013. This has largely been due to the introduction of ACTs following the resistance witnessed against chloroquine as well as an increase in the number of control measures such as the use of insecticide treated nets, long lasting insecticidal nets (LLIN), vectors surveillance and intermittent preventive treatment in pregnancy (IPTp) and implementation of the WHO policy on test, treat and track. Despite the reported decrease, most of the endemic countries across sub Saharan Africa still bear the greatest burden of the disease where 90% of the deaths are reported with more than 75% of the mortalities in children under five.

Ghana National Malaria Control Programme (GNMCP) reports reveal that in 2006 malaria accounted for 37.5% of all out patient consultations, 36.0% of all hospital admissions, and about 33.4% of all mortality in children under age five years. Following the recommendation of the WHO, Ghana changed it malaria treatment guidelines adopting artesunate and amodiaquine as first line for the treatment of uncomplicated malaria to replace chloroquine. By 2012, hospital statistics across the country revealed that malaria was responsible for 38.93% of the outpatient consultations and 38.80% of admissions. Of those admitted for malaria, 63% were children under 5 years of age while pregnant women constituted 16.8%. Furthermore, According to the Ghana Health Service (GHS) report of 2012, malaria accounted for 22.4% deaths in children less than five years of age and 3.4% deaths among pregnant women. Over the last decade, studies in Ghana have demonstrated that artesunate and amodiaquine combinations are not only efficacious in clearing the malaria parasites from patients but if used for intermittent preventive treatment programmes for children under five could effectively clear more than 90% of the parasite in this age group.

Different studies have demonstrated very high level of asymptomatic malaria parasitaemia in both less than 5 years old and school age children. In 2009, Ahorlu et al, reported a parasite prevalence of 25% in less than five year old children in the Shime sub district in the coast of Ghana. In the same light, reported a malaria parasitaemia prevalence of 58.6% among school children in the Ejusu Juaben District, while reported a 41.5% prevalence of malaria parasitaemia in Ghanaian school children in the Ashainti and Upper West regions of the country. A related study in the Dodowa area demonstrated that children with high levels of asymptomatic parasitaemia have a higher risk of coming down with clinical malaria.

The link between one parasite carrier or infected individual and the next relies on the mosquito picking up the parasite during a blood meal. This means that even if all patients with malaria are treated of the disease, those individuals who carry the parasite and are not ill could redistribute it to the healthy population with the help of the mosquito and therefore, the cycle simply continues. The high incidence of asymptomatic parasitaemia serves as a reservoir that fuels the malaria transmission cycle. If the parasite is cleared from the blood of asymptomatic individuals as well as the sick patients with the very efficacious Artemisinin-based Combination Therapy (ACT), then, even the most effective mosquito vector would have nothing to transmit following a blood meal.

Continuous exposure to the malaria parasite has led to the development of immunity, especially in adults in endemic areas. This is often a slow process as it depends on repeated exposure to the parasites. This explains why children carry the greatest burden of the disease. As they grow beyond age 5 years, the prevalence of malaria or parasitaemia in this group begins to decrease following the development of immunity to the parasite. Age, therefore, has a great role to play when looking at the dynamics of the malaria burden. A study of trends in malaria admission in a Health Centre in Cameroon has demonstrated that the variation in the prevalence of malaria effectively reflected a variation in the prevalence in children age one to less than 15 years. In endemic areas, children have been reported to harbour relatively high levels of the parasite without coming down with the disease, and the population is continuously exposed to the infected mosquitoes. That is, the already parasitised individuals can be re-infected either with the same parasite, thus, increasing the parasite load or other parasite species leading to a co-infection in areas with more than one species of Plasmodium. On the other hand, the uninfected mosquito is initially harmless even if it bites. However, it becomes infective when infected by a parasitised individual who could either be febrile or asymptomatic. Therefore, while enormous effort is being made to prevent man-vector contact through the use of treated nets, the benefits from using these nets could be amplified if such programmes integrate mass parasite clearance as part of their agenda. That is mass testing, treatment and tracking should precedes the mass distribution of LLIN in a given area or intermittent preventive treatment in children.

There has been concerted effort in the past decade to evaluate the possible effects of massive parasite clearance using intermittent preventive treatment in less than five year old children in different part of Africa with interesting results. Most studies however, focused on the clinical incidence of the disease as outcome measure which has been observed to reduce with a range of between 20-80% depending on a number of factors. In a longitudinal study in a Coastal village in Ghana, Ahorlu et al, demonstrated that associating IPTc with home based management of malaria by community workers could clear more than 90% of the parasite pool in the community. This intervention reduced malaria parasitaemia prevalence from 25% at baseline to 1% at evaluation using artesunate and amodiaquine. This low level of parasitaemia in the study population was found to persisted over a period of two years. Though, this intervention had targeted only under 5 years children, it revealed the potential role intermittent preventive treatment of the population could play in reducing malaria prevalence and consequently paving the way for malaria elimination. Given that old members of the household are likely to have some immunity to the malaria parasite, they however, represent the reservoir that refuels the parasite pool whenever it is reduced by IPTc. Therefore, for sustainability of such implementation intervention, intermittent preventive treatment would be of greater benefit if all the members of each given household are targeted for mass testing, treatment and tracking at baseline and consequent prompt home-based treatment for suspected cases. Bearing in mind that huge resources are required for IPT of whole communities, it has been suggested that mass screening of whole communities be carried out once a year while IPTc be conducted regularly in combination with the home based management. This could further enhance the efforts.

Implementation of rapid scale-up preventive interventions in the past decade has led to a reasonable decrease in the burden of the malaria (WHO 2011) especially given the introduction of the WHO policy of test, treat and track (T3) (WHO 2012). The challenges involved with translating research scenarios into implementation are enormous. It is important to understand the bottlenecks that hinder this process in order to undertake mass testing, treatment and tracking in a large scale using existing health systems, especially in an era when global funding for health services is slowing down.

Any effective control strategy that interrupts the link between man, the parasite and the vector could seriously reduce the transmission of malaria. In this light, interventions focused on clearing of the parasites in asymptomatic individuals in combination with intensive use of other control measures could pave the way for pre-elimination of the parasite in endemic communities. This study aims at reducing the asymptomatic parasitaemia in the Pakro sub district of the Eastern Region of Ghana by conducting MTTT for malaria parasitaemia among household members of age 2 months and older and carrying out targeted treatment of all cases with confirmed asymptomatic parasitaemia or clinical malaria. These interventions intend to follow up enrolled participants over a period of two years. Hospital records will also be studied to document trends in malaria admissions and occurrence of other diseases in the area before and after the interventions.

Rationale Malaria continues to poses a serious burden to the local populations in sub-Sahara Africa. Several efforts have been made to scale up interventions that work such as preventing man-vector contact, intermittent preventive therapy, seasonal malaria chemoprophylaxis as well as TTT for febrile patients. However, much still has to be done to target the mass testing, treatment and tracking of whole populations in order to reduce the parasite load before implementing the above mentioned interventions. Though SMC is adopted for selected localities in Ghana, MTTT could be used to drastically bring down the parasite load in a given population before the implementation of interventions such as SMC. Elsewhere, it has been demonstrated that incorporating the antimalarials in vaccination programmes could delay the first malaria episode in children under five. Furthermore, MTTT of children in a community in Ghana has been reported to reduce the parasite load in a given community from 25% to 1%. The questions that remain are - could this be scaled up? What proportion of the community could be covered over a given time? What would it take to accomplish MTTT in large scale? In designing interventions that aim at reducing the burden of malaria in children under five, for example, MTTT could be used to clear parasites from the general population before the interventions are implemented. This is because the adults who are not often included in the interventions that target children under 5 years old tend to act as reservoirs that fuel the transmission. To solve the problem of personnel who are limited at the level of the health service and coverage, this study will be making use of the existing network of community nurses/volunteer teams that are used during vaccination programmes. These volunteers, who recite in the communities, will carry out the interventions in the given communities and conduct the home-based management of malaria between interventions thereby increasing surveillance and reducing cost. Furthermore, to solve the problem of stock-outs and quality of the RDTs and antimalarials, the investigators will make use of SMS through mobile phones and a team will conduct monthly monitoring and evaluation of the field activities of the volunteers as well as refill the medicine and RDTs. The volunteers will be trained based on the 2014 guidelines for managing uncomplicated malaria.

The investigators hypothesize that in the Pakro sub district, there are more asymptomatic malaria cases than the symptomatic cases reported by hospital records and that if the investigators carry out MTTT in combination with home-based management of malaria in specific communities over two years, a large proportion of the parasite reservoir will be cleared and consequently open up possibilities for pre-elimination of malaria in the area. It is also intended that the bottlenecks involved in scaling up mass testing, treatment and tracking will be documented in order to facilitate the process.

Main objective The main objective of this study is to explore the impact of scaling up mass testing, treatment and tracking on malaria prevalence among children under fifteen years of age in the Pakro sub district of Ghana.

Specific Objectives

1. To evaluate the effect of scaling up targeted MTTT/home-based treatment on malaria parasitaemia and hospital consultations and admissions.
2. To determine the prevalence of asymptomatic parasitaemia among afebrile participants.
3. To reduce the burden of malaria in the participating communities.
4. To document challenges which hinder the scale up of mass testing, treatment and tracking of malaria in Ghana.
5. To conduct a cost benefit analysis of the intervention in the area.

Methodology

Study Area Pakro is one of five sub-districts in the Akwapim south district health directorate (DHD) in the Eastern region of Ghana. The Akwapim south district lies within the semi-equatorial climatic region, and experiences two rainfall seasons in a year, with an average rainfall of 125cm to 200cm. The first rainy season begins from May to June with the heaviest rainfall in June, whilst the second rainy season begins from September to October. According to the Ghana Statistical Service (GSS), the average household size in the Akwapim South district is estimated to be 4.0 whilst the average number of households per house or compound is estimated to be 1.6. The Pakro sub-district has an estimated population of 7,889, and is bounded to the east by Akwapim North district; to the north by Ayensuano district; and to the west by Nsawam Adoagyiri Municipality. The sub-district is made up of 22 communities, and has 3 health care facilities (1 Health Centre and 2 Community-Based Health Planning Service (CHPS) compounds).Due to limited resources, only seven communities will be selected for this study. This include Abeasi Newsite, Fante Town, Zongo (Adjenase/Kweitey), Piem/odumsisi, Adesa Latebibio, Sacchi/Tabankro and Odum Tokuro. These are communities with a relatively high population density. The Pakro Health Centre is one of thirty sentinel sites monitoring malaria prevalence in the country coordinated by the Noguchi Memorial Institute for Medical Research (NMIMR). Malaria parasite positivity rate was estimated to be 45.7% in 2014 (DHD, 2014). In the same year anaemia among pregnant women at 36 weeks of gestation was 21%.

Study participants

Community entry activities to sensitise the chiefs and the general population will be conducted at the beginning of the study through meetings and durbars. Once the community leaders and the population have accepted the project, the household will be numbered and participants per household will be registered during a household census. All households will be given a unique identification code. Each individual within the household will be assigned a code that links them to a particular household and community. After obtaining consent from the household heads, the children will be enrolled but individual assent and consent will be obtained from the other adolescents and adults in the household. A cohort of 460 children age 6 months to 15 years will be selected and enrolled into the longitudinal study which will consist of prevalence surveys undertaken before each MTTT. Caregivers of the children in the cohort will be enrolled for the community surveys using questionnaires. In this implementation research the entire population of the seven selected communities will be tested, treated and tracked. This is intended to clear the parasite pool in the community.

Intermittent preventive treatment for the household members

The research team together with Community assistants/volunteers will conduct house-to-house testing (using RDTs) of all children (from 6 months old) and adults residing in 7 selected communities for the presence of malaria parasites. For this study, the investigators will use the Ag P.f RDT which detects histidinie-rich proteins II antigens (HRP-2 Ag) specific to P. falciparum in human blood. The RDTs will be supplied by the Ghana Health service through the National malaria control programme which uses the services of WHO-FIND Lot Testing Programme for quality assurance. Thus, the investigators are using the same RDT that has been procured by the NMCP and are being used routinely in Ghana. To enable follow up studies in a case where treatment failure is reported, 200ul (two drops) of blood will be collected on filter paper. This will be used to determine immunological parameters such as antibody levels to specific antigens using Polymerase Chain Reaction (PCR) and Enzyme Linked Immunosorbent Assay (ELISA). RDT confirmed cases who are treated but presents persistent malaria related symptoms such as fever on day 7 will be tested using microscopy and to determine clinical failure. This study is not designed to test for parasite resistance to drug (drug efficacy) and the Project clinicians will advise on the next line of action. This could be taken up by a masters' student. However, the student will need to submit a different protocol to the ERC for approval). All participants confirmed (using RDTs) to be carrying the malaria parasite will be treated using ACTs following the Ghana National Malaria Treatment Guidelines and followed up on days 1, 2, 3 during treatment as DOTs (Directly observed therapy) and on day 7 post treatment. The research team together with Community volunteers will be provided the treatment guidelines which specify the dosage for each treatment regimen. Participants who receive the treatment will be observed for five minutes to ensure that they retain the drug. Those who vomit within this period will have the treatment repeated.

Follow-Up

All treated cases will be followed up on days 1, 2, 3 during treatment and day 7 post-treatment to ensure that the participants take the drugs on time as well as document and report all adverse effects.

Questionnaire/Focus group Discussion

The questionnaire will include questions about malaria treatment, prevention and control measures practiced by the household members. Occupants of the household will provide a blood sample for testing. Focus group discussions will be organized with community members and health care workers to increase the scope of information obtained.

Timely treatment of suspected febrile malaria case in the community

In other to render operational the home-based management component of the project, two volunteers will be selected from each community and trained on home-based management of malaria and be provided with the protocol, RDTs and ACTs. The interventions will be carried out quarterly (see the timetable). Between one MTTT intervention and the next trained community members will provide prompt home-based treatment for children and adults reporting signs and symptoms of malaria and confirmed to be carrying the parasite using RDTs. This will be done using national malaria management protocol. There will be monthly visits by the research team to supervise the community volunteers involved in home-based management to ensure that the protocol is being respected as well as replenish their stocks. There is a need to visit the health facilities that service the community to enable tracking and linking of medical records with study participants (a master student is required for this component). The investigators hypothesize that a reduction in parasite load in the community will consequently lead to a reduction in the number of hospital malaria related consultations and admissions paving the way for pre-elimination. This will be realised by comparing baseline hospital malaria admission data to evaluation data. MTTT has already been adopted by the NMCP as one of the control and elimination activities and the investigators are anticipating its being scaled-up in the country, and therefore documenting its implementation challenges will inform the decision in the future.

Sample size

This is an implementation study aimed at enrolling an entire population estimated at 4500 participants from the 7 selected communities in Pakro sub district. This population was obtained following data from a head count in preparation for the mass distribution of LLIN in 2016 - Abase newsite = 800, Fante town = 1450, Adjenase/Kwettey = 1102, Piem/Odumsisi = 323, Adesa/Nsuablaso = 480, Sacchi/Tabnkro = 201, Odumtokro = 129 (Pakro Health Centre records). However, since the target effect of this intervention is focused at the children age 6 months to 15 years, a community survey with a sample of 368 children will be needed to determine the malaria prevalence projected at 50% in the study population. This has been determined using the formula of Yamane where n = N/[1+N(е)2] (Israel 1992) considering a 95% confident level (CI) and ±5% precision. Assuming a loss to follow up of 10% and a non-response rate of 10%, the sample size is readjusted to 460 children calculated from (38/1-0.2) for the community survey. At evaluation the available sample size will be determined. This is the group for which questionnaires will be administered. Following a census of the households, children under 6 months to 15 years old will be randomly selected for the longitudinal cohort study, they will then be divided into the various age groups 6 months to 11 months, 1-4 years, 5 -10 years and 11-15 years. For each age group the investigators will randomly select 116 children.

Data collection

Following consent, blood will be drawn from a finger prick. All participants will be tested for the presence of malaria parasites using RDTs. Additionally, blood will be collected on filter paper to enable molecular characterization in case treatment failure is observed in a given patients as explained above. All samples will be stored at NMIMR. To test for anaemia (for children in the cohort study only), a portable automated Hemocue photometer will be used to determine the concentration of Haemoglobin. Anaemia in this study is defined as Hb levels less than 10g/dl. Children with severe anaemia (Hb less than 7g/dl) will be referred to the Pakro Health Centre for follow up. At evaluation, family members will be asked questions on how much they used to spend on malaria before the intervention and how much they have spent after. Malaria case management records before and after the intervention will be consulted, firstly to determine the change in prevalence and also for cost benefit analysis purposes.

Data Management and Analysis

Data Management will be conducted with the support of the Data management unit in the Department of Epidemiology of NMIMR. A database will be created to manage the data. Data will be entered into Epi-info and analysed using SPSS. The unit of enrollment will be the household. Malaria prevalence will be reported as, proportion of subjects identified during the study period with RDT confirmed clinical malaria with temperature ≥37.5 or asymptomatic parasitaemia and stratified by subject characteristics, including age, sex and community. A Chi square statistic will be used to compare prevalence across age and gender categories as well as communities. To determine whether interventions had an effect on the prevalence of malaria in the area, the baseline prevalence data will be compared with the evaluation data. Also a cost benefit analysis will be conducted by comparing what the NMCP put in in previous years to treat malaria to what it would spend if MTTT is implemented.

Problems Anticipated

It is anticipated that ACTs and RDTs supplies could delay. In order to avoid this, the investigators have approached the national malaria control programme to arrange for drugs and RDTs supply through the Eastern Regional Store. The investigators anticipate the number allocated to houses in the communities could be wiped and so the data for each house is linked to the name of the house. This could enable easy tracing of the participants. In the field the investigators will use forms that already carry the names of the families following the census. Names of new people could be added.

Project Management

The PI will carry out day to day implementation and supervise of all aspect of the project. Co-PIs are part of the implementation team and will participate in the decision making at all stages of the project. The Research assistant will help in facilitating project logistics. The Regional/District Health Directorates through the health facility in Pakro will facilitate the work. The volunteers are community members that assist in data collection while the driver facilitates movements.

Quality Assurance

In order to ensure the quality of data collected, 20 volunteers will be trained and 14 will be selected for the project. The questionnaires will be pretested and corrections effected. All data collected will be cross checked by two persons in the fields. To avoid loss of data, all data from the field will be recorded in the data transfer sheet before being transferred to the data management unit. All ACTs and RDTs will be procured from the National Malaria Programme through the Eastern Region medical store. The expiry dates for all procurements made will be verified.

Ethical Consideration

The ethical clearance for this study will be sought from the NMIMR-IRB

Consent Procedure

The investigators will obtain consent at different levels. Administrative authorization will be obtained from the Ghana Health Service. There will be community consent given by the chiefs, households consent given by the head or parents/caretakers for children below 18 years, individual assent for 12-17 years old and consent for adults in each household. People from 18 years old are considered as Adults.

Privacy and confidentiality

All information/samples obtained from participants and their results will be kept confidential and not be released to a third party.

Data storage and Usage

This information will be stored in a secure location at the Epidemiology Department of NMIMR. Some staff of Epidemiology Department of NMIMR may access the data for research purposes only, such as malaria prevalence studies in asymptomatic individuals. Findings will be published with no reference to any personal identifiers. The data collected will be stored for a period of five years at NMIMR.

Data ownership

Data resulting from this study is own by the NMIMR.

Risk

There is no health threatening risk. Some participants may vomit within five minutes after taking the ACTs. It is assumed that if a patient vomits within five minutes he/she has not absorbed an acceptable quantity of the medicine. In this case the treatment will be repeated. Some other patients may show adverse reactions after taking the drugs such as stomach upset, dizziness, nausea, body weakness, etc. In other to cross check for some of these adverse events, the team will monitor volunteers for four days following treatment.

Conflict of Interest

The PI and co-PIs declare no conflict of interest in the execution of this project.

Benefits

All confirmed malaria parasitaemia cases will be treated for free. Continuous monitoring and treatment of confirmed cases will improve the health of residents. The study will reduce household spending on malaria thereby free some funds to be spent on other household items. This project could reduce the malaria related burden in the implementing communities.

ELIGIBILITY:
Inclusion Criteria:

1. Overall inclusion criteria for MTTT:

   * Be aged 2 months or older
   * Be resident in the study area
   * Have completed and signed the consent for adults or assent form for children 12-17 years.
2. Inclusion Criteria for children in the cohort study:

   * Be age range 6 months to 14 years
   * Be resident in the study area for the period of the study.
   * Be willing to participate
   * Parent or guardian have completed and signed consent form

Exclusion Criteria:

* If an individual intents to stay less than one year in the study site
* Be absent at some time because he/she is schooling in a boarding school
* Has a life threatening illness (excluding malaria).

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The rate of asymptomatic malaria parasitaemia among afebrile children aged 6 months to 15 years and adults in the Pakro sub district will be known. | Once every 4 months, over a period of 24 months
  The change in the rate of asymptomatic parasistaemia at evaluation compared to baseline. This will be determined by testing for the presence of malaria parasite in healthy participants without a history of fever in the last 48 hours before an intervention. This will be done using rapid diagnostic test. The temperature will be taken before the the test to ensure that the patients are not febrile. Questionnaires will be used to collect data on the prevalence of febrile illnesses.
The proportion hospital admissions due to malaria that are averted as a result of MTTT implementation will be determined. | 24 months
  The effect of MTTT on hospital admissions in the intervention communities will be evaluated by comparing the proportion of confirmed malaria cases during the MTTT intervention period to the proportion of confirmed malaria cases period before implementation of the MTTT intervention at the Pakro Health Centre. Data on malaria test results will be collected from hospital registers. The proportion will be defined as (number of confirmed malaria cases/number of participants tested for malaria) *100. Questionnaires, focus group discussions and In-depth interviews will be used to gather complementary information to obtain a holistic picture of the effect of the interventions in the community.
The list of challenges that needs to be addressed to enable scale-up of MTTT interventions feasible in Ghana. | 24 months
  This outcome will provide a list of challenges faced by the investigators during the implementation of MTTT. It will also state how many challenges were addressed and at what level. A detailed description will be made of how each challenge was addressed at the level of the community, administration and stakeholders. Data will be collected from field notes taken during monthly monitoring visits, field reports, interviews and focus group discussion.

SECONDARY OUTCOMES:
The cost benefit analysis of the scaling up MTTT intervention in the area will be known. | 24 Months
  This outcome describes the benefit in terms of number of cases of malaria prevented or amount of income saved by the participants or resources saved by the health system as a result of implementing MTTT

CONTACTS AND LOCATIONS:
Overall Officials: Ignatius C Ndong, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Noguchi Memorial Institute for Medical Research, Accra, Greater, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from this study is own by the NMIMR. The findings of the study will be shared with the local communities, data will be published in open access journals
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2017-2019
Access Criteria: The findings of this study will be published in open access journal and the data will be made available to individual researchers upon request.

REFERENCES:
- [Background] Ahorlu CK, Koram KA, Seake-Kwawu A, Weiss MG. Two-year evaluation of Intermittent Preventive Treatment for Children (IPTc) combined with timely home treatment for malaria control in Ghana. Malar J. 2011 May 15;10:127. doi: 10.1186/1475-2875-10-127. PMID 21569634
- [Background] Ahorlu CK, Koram KA, Seakey AK, Weiss MG. Effectiveness of combined intermittent preventive treatment for children and timely home treatment for malaria control. Malar J. 2009 Dec 11;8:292. doi: 10.1186/1475-2875-8-292. PMID 20003357
- [Background] Appawu MA, Baffoe-Wilmot A, Afari EA, Nkrumah FK, Petrarca V. Species composition and inversion polymorphism of the Anopheles gambiae complex in some sites of Ghana, west Africa. Acta Trop. 1994 Feb;56(1):15-23. doi: 10.1016/0001-706x(94)90036-1. PMID 8203292
- [Background] Bousema T, Okell L, Felger I, Drakeley C. Asymptomatic malaria infections: detectability, transmissibility and public health relevance. Nat Rev Microbiol. 2014 Dec;12(12):833-40. doi: 10.1038/nrmicro3364. Epub 2014 Oct 20. PMID 25329408
- [Background] Bull PC, Lowe BS, Kortok M, Molyneux CS, Newbold CI, Marsh K. Parasite antigens on the infected red cell surface are targets for naturally acquired immunity to malaria. Nat Med. 1998 Mar;4(3):358-60. doi: 10.1038/nm0398-358. PMID 9500614
- [Background] Dicko A, Sagara I, Sissoko MS, Guindo O, Diallo AI, Kone M, Toure OB, Sacko M, Doumbo OK. Impact of intermittent preventive treatment with sulphadoxine-pyrimethamine targeting the transmission season on the incidence of clinical malaria in children in Mali. Malar J. 2008 Jul 8;7:123. doi: 10.1186/1475-2875-7-123. PMID 18611271
- [Background] Koram K, Quaye L, Abuaku B. Efficacy of amodiaquine/artesunate combination therapy for uncomplicated malaria in children under five years in ghana. Ghana Med J. 2008 Jun;42(2):55-60. PMID 19180204
- [Background] Kweku M, Webster J, Adjuik M, Abudey S, Greenwood B, Chandramohan D. Options for the delivery of intermittent preventive treatment for malaria to children: a community randomised trial. PLoS One. 2009 Sep 30;4(9):e7256. doi: 10.1371/journal.pone.0007256. PMID 19789648
- [Background] Ndong IC, van Reenen M, Boakye DA, Mbacham WF, Grobler AF. Trends in malaria admissions at the Mbakong Health Centre of the North West Region of Cameroon: a retrospective study. Malar J. 2014 Aug 22;13:328. doi: 10.1186/1475-2875-13-328. PMID 25145498
- [Background] Newell K, Kiggundu V, Ouma J, Baghendage E, Kiwanuka N, Gray R, Serwadda D, Hobbs CV, Healy SA, Quinn TC, Reynolds SJ. Longitudinal household surveillance for malaria in Rakai, Uganda. Malar J. 2016 Feb 9;15:77. doi: 10.1186/s12936-016-1128-6. PMID 26861943
- [Background] Ofosu-Okyere A, Mackinnon MJ, Sowa MP, Koram KA, Nkrumah F, Osei YD, Hill WG, Wilson MD, Arnot DE. Novel Plasmodium falciparum clones and rising clone multiplicities are associated with the increase in malaria morbidity in Ghanaian children during the transition into the high transmission season. Parasitology. 2001 Aug;123(Pt 2):113-23. doi: 10.1017/s0031182001008162. PMID 11510676
- [Background] Rao VB, Schellenberg D, Ghani AC. Overcoming health systems barriers to successful malaria treatment. Trends Parasitol. 2013 Apr;29(4):164-80. doi: 10.1016/j.pt.2013.01.005. Epub 2013 Feb 14. PMID 23415933
- [Background] Sarpong N, Owusu-Dabo E, Kreuels B, Fobil JN, Segbaya S, Amoyaw F, Hahn A, Kruppa T, May J. Prevalence of malaria parasitaemia in school children from two districts of Ghana earmarked for indoor residual spraying: a cross-sectional study. Malar J. 2015 Jun 25;14:260. doi: 10.1186/s12936-015-0772-6. PMID 26109461
- [Background] Sinclair D, Zani B, Donegan S, Olliaro P, Garner P. Artemisinin-based combination therapy for treating uncomplicated malaria. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD007483. doi: 10.1002/14651858.CD007483.pub2. PMID 19588433
- [Background] Farnert A, Snounou G, Rooth I, Bjorkman A. Daily dynamics of Plasmodium falciparum subpopulations in asymptomatic children in a holoendemic area. Am J Trop Med Hyg. 1997 May;56(5):538-47. doi: 10.4269/ajtmh.1997.56.538. PMID 9180605
- [Background] WORLD HEALTH ORGANISATION Roll Back Malaria Report. Geneva: WHO; 2003. http://www.rollbackmalaria.org/microsites/wmd2011/amr_toc.html. Accessed 15 November. 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2009. Geneva: WHO; 2009 http://www.who.int/malaria/world_malaria_report_2014/en. Accessed 3 December. 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2010. Geneva: WHO; 2010. http://www.who.int/malaria/world_malaria_report_2010/en. Accessed 1 December 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2011. Geneva: WHO; 2013 http://www.who.int/malaria/publications/world_malaria_report_2013/en. Accessed 2 December 2016
- [Background] WORLD HEALTH ORGANISATION. World Malaria Report 2014. Geneva: WHO; 2014 http://www.who.int/malaria/publications/world_malaria_report_2014/en. Accessed 1 December, 2016
- [Background] WORLD HEALTH ORGANISATION (2012).
- [Background] OTUPIRI, E., YAR, D. & HINDIN, J. 2012. Prevalence of Parasitaemia, Anaemia and treatment outcomes of Malaria among School Children in a Rural Community in Ghana. Journal of Science and Technology (Ghana), 32, 1-10.
- [Background] ISRAEL, G. D. 1992. Determining sample size, University of Florida Cooperative Extension Service, Institute of Food and Agriculture Sciences, EDIS.
- [Background] GHANA STATISITCAL SERVICE, 2010. Population and Housing Sensus. District Analytic Report: Akwapim South District.
- [Background] GNMCP 2006. Ghana National Malaria Control Programme: Ghana Health Service Report 2006 Accra.
- [Background] DISTRICT HEALTH DIRECTORATE, 2015. District Annual Report 2015, Akwapim South, Aburi, Ghana
- [Background] DISTRICT HEALTH DIRECTORATE, 2014. District Annual Report 2014, Akwapim South, Aburi, Ghana.
- [Result] Ndong IC, Okyere D, Enos JY, Amambua-Ngwa A, Merle CSC, Nyarko A, Koram KA, Ahorlu CS. Challenges and perceptions of implementing mass testing, treatment and tracking in malaria control: a qualitative study in Pakro sub-district of Ghana. BMC Public Health. 2019 Jun 6;19(1):695. doi: 10.1186/s12889-019-7037-1. PMID 31170964
- [Derived] Ndong IC, Okyere D, Enos JY, Mensah BA, Nyarko A, Abuaku B, Amambua-Ngwa A, Merle CSC, Koram KA, Ahorlu CS. Prevalence of asymptomatic malaria parasitaemia following mass testing and treatment in Pakro sub-district of Ghana. BMC Public Health. 2019 Dec 3;19(1):1622. doi: 10.1186/s12889-019-7986-4. PMID 31795981

DOCUMENTS (4):
  • Study Protocol (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04167566/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Anlysis Plan (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04167566/SAP_001.pdf
  • Informed Consent Form (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04167566/ICF_002.pdf
  • Statistical Analysis Plan: results (2019-03-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04167566/SAP_003.pdf